CLINICAL TRIAL: NCT04546178
Title: Implementation and Evaluation of Prolonged Exposure Psychotherapy for Adverse Events in Early Phase Psychosis With Comorbid Substance Misuse
Brief Title: Psychotherapy for Psychosis, Adverse Events, and Substance Misuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Queen Elizabeth II Health Sciences Centre Foundation (Unknown); Research Nova Scotia (Unknown); Killam Laureates (Unknown)
Responsible Party: Principal Investigator, Victoria Patterson, Principal Investigator, Dalhousie University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: REB1025608
Record Dates: First submitted 2020-08-28; First posted 2020-09-11 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Psychotic Disorders; Stress Disorders, Traumatic; Substance Use
Keywords: Substance misuse; Schizophrenia spectrum disorders; Adversity; Cognitive Behavioral Therapy (CBT)
MeSH Terms: conditions — Psychotic Disorders; Stress Disorders, Traumatic; Substance-Related Disorders | interventions — Therapeutics; Antipsychotic Agents

STUDY DESIGN:
Intervention Model Description: A single-case experimental design (SCED), specifically, a multiple-baseline design (MBD; Kratochwill et al., 2010) will be used; the MBD temporally staggers intervention start times across participants, thereby creating a control group composed of each individual's pre-intervention scores. Randomization of each participant's treatment start time will be used to increase internal validity and minimize bias (Kratochwill & Levin, 2010). Participants will be randomized using a random sampling/assignment generator (randomizer.org). An MBD is an ideal design for a study focused on the optimization of PE+ and this approach will allow a fine-grained assessment (Lobo et al., 2017) of its effectiveness in EPP. This design can also detect significant changes during each phase of the intervention. In order to meet standards of evidence for SCEDs, this study will include a total of five treatment phases, which exceeds the recommended minimum of three phases (Kratochwill et al., 2010).
Who Masked: Outcomes Assessor
Masking Description: The trained therapist conducting the symptom assessments will not have access to information regarding that participant's treatment, and the person providing the treatment will not have access to the information regarding assessments of that participant's symptoms. Therapists will only conduct a symptom assessment for participants that are working with another therapist; they may not conduct a symptom assessment for participants with whom they are working through the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PE+ intervention group (Experimental): This group will participate in 15 sessions of PE+ therapy and participate in frequent symptom assessments; this is the same group of participants as the pre-intervention scores group, but they have crossed over from pre-intervention phase into intervention (active) phase.
  Interventions: Behavioral: Prolonged exposure (PE)+ therapy; Other: Treatment as usual (TAU)
- Pre-intervention scores group (TAU) (Active Comparator): This group will participate in symptom assessments but will not receive the PE+ intervention until the begin the active part of the trial. Participants in this group have been diagnosed with a psychotic disorder, have also experienced adversity, and use substances. This group will receive medication for psychosis as well as access to standard education programs and clinical care; thus treatment as usual (TAU).
  Interventions: Other: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Prolonged exposure (PE)+ therapy — The intervention will be adapted prolonged exposure therapy, called PE+ therapy. Participants will receive 15 weekly 90-minute sessions of PE+; these appointments will be divided into five sets of three sessions each: 1) psychoeducation about AEs, SM, and the interplay of both with psychosis; 2) emotion regulation strategies; 3) imaginal exposures, 4) in vivo exposures, and 5) review of treatment and planning for termination and maintenance.
  Other Names: PE+ therapy
  Arms: PE+ intervention group
Other: Treatment as usual (TAU) — The intervention will be antipsychotics prescribed by clinicians working within the Nova Scotia Early Psychosis Program (NSEPP) as well as case management supplied by their primary nurse. Program participants will have access to educational programs about psychosis, skills/vocational training, as well as familial education and support.
  Other Names: Antipsychotics and program access

SUMMARY:
People with psychosis have significantly higher rates of adversity (e.g., abuse) and substance misuse (i.e., problematic drug and alcohol use) than people with other mental illnesses. Research has found that adversity and substance use both negatively influence recovery from a psychotic disorder. Currently, there are few treatment options for people living with psychosis, substance misuse, and adversity-related symptoms (e.g., anxiety, depression). This is especially true for young adults who are in the first years of a psychotic illness (i.e., early phase psychosis; EPP) who may be in the best position to benefit from treatment because they have not been ill for as long as others with more chronic psychosis (i.e., >10 years). Research has demonstrated that Prolonged Exposure (PE), a psychological therapy that helps improve adversity-related symptoms, may be appropriate for people in EPP, although there is limited evidence regarding its adaptation from use in chronic psychosis to EPP. The aim of the proposed study is to adapt and optimize PE therapy for young adults in EPP. We aim to recruit 20 individuals from the Nova Scotia Early Psychosis Program (NSEPP) aged 19-35 who will participate in 15 sessions of adapted PE; we will compare their scores before and after treatment on measures of psychotic symptoms, amount and frequency of substance use, and adversity-related problems. Our goal is to target two factors that may be contributing to and maintaining negative outcomes: avoidance and hopelessness. These factors will be addressed by asking participants to face feared reminders of adversity and learn new ways to think about adverse experiences and mental health problems. The adaptation and application of this evidence-based intervention has the potential to create a new treatment avenue for EPP, reducing impairment and distress, and improving recovery rates.

ELIGIBILITY:
Inclusion Criteria:

* Current patient at the Nova Scotia Early Psychosis Program (NSEPP) for the duration of the study
* Aged 19-35 years
* Diagnosis of a primary psychotic disorder (i.e., schizotypal disorder, delusional disorder, brief psychotic disorder, schizophreniform disorder, schizophrenia, schizoaffective disorder, substance/medication-induced psychotic disorder, other specified schizophrenia spectrum and other psychotic disorder, unspecified schizophrenia spectrum and other psychotic disorder)
* Diagnosis of a primary psychotic disorder within the past 5 years; participants must not surpass this 5-year diagnostic window whilst enrolled in the study
* Have experienced 1 or more negative, distressing lifetime adverse events (e.g., child abuse, discrimination) listed on the Trauma and Life Events (TALE) checklist that the participant indicates still affects them now
* At least one score within the "moderate" or "high" risk range for any substance (except tobacco products) on the WHO Alcohol, Smoking and Substance Involvement Screening Test (ASSIST)
* Speaks and understands English

Exclusion Criteria:

* Aged 36 and older
* Aged 18 and younger
* Score in the 'high risk' range for cocaine use on the ASSIST
* Participant does not speak or understand English
* Current involuntary inpatient admission in a hospital or under a Community Treatment Order
* Documented, diagnosed intellectual disability (ID)
* Not currently participating in any intervention designed to reduce substance use or treat symptoms related to adverse events (e.g., PTSD)

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Beck Hopelessness Scale (BHS); Change in hopelessness | Study weeks 1, 2; depending on randomization to intervention start time: administered weeks 3 through 20, 8 weeks following study week 18,19, or 20, and 9 weeks following study week 18,19, or 20 (see description above for more detail)
  This 20-item true/false scale measures hopelessness in participants; we will use the total score on this measure as an indicator of hopelessness. Scores range from 0 to 20; higher scores indicate greater hopelessness.
  Detailed timeline: Pre-intervention baseline assessment (study week 1); pre-intervention follow-up appointments (study weeks 2; 2,3; or 2,3, and 4; depending on randomization); pre-intervention assessment 1 (study week 3,4, or 5, depending on randomization); intra-intervention assessment 2 (study week 6,7, or 8, depending on randomization); intra-intervention assessment 3 (study week 9,10, or 11, depending on randomization); intra-intervention assessment 4 (study week 12,13, or 14, depending on randomization); intra-intervention assessment 5 (study week 15,16, or 17, depending on randomization); intra-intervention assessment 6 (study week 18,19, or 20, depending on randomization); 8 weeks post-assessment 6 (week 18, 19, or 20); 9 weeks post-assessment 6
Brief Experiential Avoidance Questionnaire (BEAQ); Change in avoidance | Study weeks 1, 2; depending on randomization to intervention start time: administered weeks 3 through 20, 8 weeks following study week 18,19, or 20, and 9 weeks following study week 18,19, or 20 (see description above for more detail)
  This 15-item scale measures avoidance in participants; we will use the overall score on this measure as an indicator of avoidance. Scores range from 15 to 90; higher scores indicate greater avoidance.
  Detailed timeline: Pre-intervention baseline assessment (study week 1); pre-intervention follow-up appointments (study weeks 2; 2,3; or 2,3, and 4; depending on randomization); pre-intervention assessment 1 (study week 3,4, or 5, depending on randomization); intra-intervention assessment 2 (study week 6,7, or 8, depending on randomization); intra-intervention assessment 3 (study week 9,10, or 11, depending on randomization); intra-intervention assessment 4 (study week 12,13, or 14, depending on randomization); intra-intervention assessment 5 (study week 15,16, or 17, depending on randomization); intra-intervention assessment 6 (study week 18,19, or 20, depending on randomization); 8 weeks post-assessment 6 (week 18, 19, or 20); 9 weeks post-assessment 6 (week 18, 19, or 20)
World Health Organization's Alcohol, Smoking, and Substance Involvement Screening Test (WHO ASSIST); Change in substance use | Eligibility assessment (week 0); Depending on randomization to intervention start time: administered weeks 3 through 20, 8 weeks following study week 18,19, or 20, and 9 weeks following study week 18,19, or 20 (see description above for more detail)
  The ASSIST measures substance use; we will use the total score for each substance as an indicator of substance use. Scores range from 0-39 for each subscale; higher scores indicate substance misuse.
  Detailed timeline: Eligibility screening assessment (pre-study enrollment); pre-intervention assessment 1 (study week 3,4, or 5, depending on randomization); intra-intervention assessment 2 (study week 6,7, or 8, depending on randomization); intra-intervention assessment 3 (study week 9,10, or 11, depending on randomization); intra-intervention assessment 4 (study week 12,13, or 14, depending on randomization); intra-intervention assessment 5 (study week 15,16, or 17, depending on randomization); intra-intervention assessment 6 (study week 18,19, or 20, depending on randomization); 8 weeks post-assessment 6 (week 18, 19, or 20); 9 weeks post-assessment 6
Positive and Negative Syndrome Scale (PANSS) - Negative subscale; Change in negative psychotic symptoms | Study week 1; pre-intervention assessment 1 (study week 3,4, or 5, depending on randomization); 8 weeks following study week 18,19, or 20 and 9 weeks post study week 18,19, or 20 (depending on randomization to intervention start time)
  The PANSS measures positive and negative psychotic symptoms; we will use the total score of the negative symptoms subscale on this measure as an indicator of negative symptoms. Scores range from 7 to 49; higher scores indicate greater negative symptoms.
Social and Occupational Functioning Assessment Scale (SOFAS); Change in functioning | Study weeks 1, 2; depending on randomization to intervention start time: administered weeks 3 through 20, 8 weeks following study week 18,19, or 20, and 9 weeks following study week 18,19, or 20 (see description above for more detail)
  This clinician-reported instrument measures social and occupational functioning. Scores on this measure range from 1 to 100; higher scores indicate greater functioning, lower scores indicate greater impairment in functioning.
  Detailed timeline: Pre-intervention follow-up appointments (study weeks 2; 2 and 3; or 2,3, and 4; depending on randomization to intervention start time); pre-intervention assessment 1 (study week 3,4, or 5, depending on randomization); intra-intervention assessment 2 (study week 6,7, or 8, depending on randomization); intra-intervention assessment 3 (study week 9,10, or 11, depending on randomization); intra-intervention assessment 4 (study week 12,13, or 14, depending on randomization); intra-intervention assessment 5 (study week 15,16, or 17, depending on randomization); intra-intervention assessment 6 (study week 18,19, or 20, depending on randomization); 8 weeks post-assessment 6 (week 18, 19, or 20); 9 weeks post-assessment 6 (week 18, 19, or 20)

SECONDARY OUTCOMES:
Trauma Symptom Checklist-40 (TSC-40); Change in adversity sequelae | Study weeks 1, 2; depending on randomization to intervention start time: administered weeks 3 through 20, 8 weeks following study week 18,19, or 20, and 9 weeks following study week 18,19, or 20 (see description above for more detail)
  TSC-40 measures adversity sequelae. We will use the total score and the subscale scores (e.g., dissociation, anxiety, depression). Total scores range from 0 to 120; higher scores indicate greater psychopathology.
  Detailed timeline: Pre-intervention baseline assessment (study week 1); pre-intervention follow-up appointments (study weeks 2; 2,3; or 2,3, and 4; depending on randomization to intervention start time); pre-intervention assessment 1 (study week 3,4, or 5, depending on randomization); intra-intervention assessment 2 (study week 6,7, or 8, depending on randomization); intra-intervention assessment 3 (study week 9,10, or 11, depending on randomization); intra-intervention assessment 4 (study week 12,13, or 14, depending on randomization); intra-intervention assessment 5 (study week 15,16, or 17, depending on randomization); intra-intervention assessment 6 (study week 18,19, or 20, depending on randomization); 8 weeks post-assessment 6; 9 weeks post-assessment 6
Positive and Negative Syndrome Scale (PANSS) - Positive subscale; Change in positive psychotic symptoms | Study week 1; pre-intervention assessment 1 (study week 3,4, or 5, depending on randomization); 8 weeks following study week 18,19, or 20 and 9 weeks post study week 18, 19, or 20 (depending on randomization to intervention start time)
  The PANSS measures positive and negative psychotic symptoms; we will use the total score of the positive symptoms subscale on this measure. Scores range from 7 to 49; higher scores indicate greater positive symptoms.
Clinical Global Impression - Severity of Illness and Improvement of Illness (CGI-S & -I); Change in functioning | Study week 1; depending on randomization to intervention start time: administered 8 weeks following study week 18,19, or 20, and 9 weeks following study week 18,19, or 20 (see description above for more detail)
  The CGI-S measures the clinician's judgement of the severity of the participant's mental illness at this time and the CGI-I measures the degree of improvement from baseline; we will use the total severity score of the CGI-S and the total improvement score of the CGI-I. CGI-I scores range from 1 (Very much improved) to 7 (Very much worse); higher scores indicate worsening, lower scores indicate improvement. CGI-S scores range from 1 (Normal, not ill at all) to 7 (Among the most extremely ill); higher scores indicate greater illness severity, lower scores indicate low severity.
  Detailed timeline: Pre-intervention baseline assessment (study week 1); 8 weeks post-intervention session 15; 9 weeks post-intervention session 15
PTSD Checklist for DSM-5 - 8-item screener version | Study weeks 1, 2; depending on randomization to intervention start time: administered weeks 3 through 20, 8 weeks following study week 18,19, or 20, and 9 weeks following study week 18,19, or 20 (see description above for more detail)
  The 8-item PTSD Checklist-5 (PCL-5) will collect information about symptoms commonly associated with adversity, such as intrusive thoughts, avoidance of event reminders, loss of interest, etc. All items are on a 5-point scale ranging from "Not at all" to "Extremely"; higher scores suggest greater symptom severity. This questionnaire has previously been validated for use with individuals with psychosis.
  Detailed timeline: Pre-intervention baseline assessment (study week 1); pre-intervention follow-up appointments (study weeks 2; 2,3; or 2,3, and 4; depending on intervention start time); pre-intervention assessment 1 (study week 3,4, or 5); intra-intervention assessment 2 (study week 6,7, or 8); intra-intervention assessment 3 (study week 9,10, or 11); intra-intervention assessment 4 (study week 12,13, or 14); intra-intervention assessment 5 (study week 15,16, or 17); intra-intervention assessment 6 (study week 18,19, or 20); 8 weeks post-assessment 6; 9 weeks post-assessment 6

OTHER OUTCOMES:
Session rating scale Version 3 (SRS V3); Change in therapeutic alliance | Depending on randomization to intervention start time, this measure is administered after each intervention session; meaning it is administered through study weeks 4 to 18; 5 to 19; or 6 to 20.
  The SRS is a measure of therapeutic alliance. This instrument measures the therapeutic relationship, goals and topics covered in session, therapist approach/method, and the therapy session overall for each therapy session. This information will allow us to assess the impact of therapeutic alliance on symptom change. Participants will fill out this form following each therapy session and will place it in a sealed envelope; therapists will not have access to this information. Total scores range from 0 to 40; higher scores indicate greater therapeutic alliance and lower scores indicate problems in one or more areas of session therapeutic alliance.
Trauma and Life Events (TALE) checklist; Change in measurement of how much someone is affected by an adverse event | Eligibility assessment, 8 weeks post-assessment 6 (follow-up assessment 1).
  o This 21-item yes/no scale asks participants which of the listed events they have experienced in their lifetime (e.g., sexual abuse, traumatic entry into care). It also asks participants if any of the events they have experienced occurred more than once, and at what age(s) the event(s) occurred. This questionnaire also asks the participant whether those adverse events are affecting them now in any way. Two scores can be formed from this measure: 1) the total number of lifetime adverse events (ranging from 0-20) and 2) how much participants are currently affected by these events (0, "not at all" to 10, "extremely").

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Patterson, PhD student, Principal Investigator — Dalhousie University
Locations (1):
- Nova Scotia Early Psychosis Program (NSEPP), Abbie J. Lane Memorial Building, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patterson VC, Tibbo PG, Stewart SH, Town J, Crocker CE, Ursuliak Z, Lee S, Morrison J, Abidi S, Dempster K, Alexiadis M, Henderson N, Pencer A. Outcomes of an adapted prolonged exposure psychotherapy for people with early phase psychosis, substance misuse, and a history of adversity: the PE + trial. BMC Psychiatry. 2024 Oct 14;24(1):684. doi: 10.1186/s12888-024-06050-1. PMID 39402517
- [Derived] Patterson VC, Tibbo PG, Stewart SH, Town J, Crocker CE, Ursuliak Z, Lee S, Morrison J, Abidi S, Dempster K, Alexiadis M, Henderson N, Pencer A. A multiple baseline trial of adapted prolonged exposure psychotherapy for individuals with early phase psychosis, comorbid substance misuse, and a history of adversity: A study protocol. Front Psychol. 2022 Dec 12;13:1012776. doi: 10.3389/fpsyg.2022.1012776. eCollection 2022. PMID 36578677

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-26): https://cdn.clinicaltrials.gov/large-docs/78/NCT04546178/Prot_SAP_003.pdf